CLINICAL TRIAL: NCT03321357
Title: Test-retest-reliability and At-home-assessment Feasibility of the Five-repetition Sit-to-stand Test (5R-STS)
Brief Title: Retest-reliability and At-home-assessment Feasibility of the 5R-STS
Acronym: 5RSTS-2
Status: Completed | Type: Observational
Sponsor: Bergman Clinics (Other)
Responsible Party: Principal Investigator, Marc Schröder, MD, PhD, Bergman Clinics
Other Study IDs: 5R-STS-2
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spondylosis; Herniated Nucleus Pulposus; Spinal Stenosis Lumbar; Spinal Diseases; Spinal Instability
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spondylosis; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: five-repetition sit-to-stand test — An armless chair with a hard seat was stabilised by placing it against a wall. Seated participants were asked to come forward on the chair seat until the feet were flat on the floor and to fold their upper limbs across the chest. Participants were then instructed to stand up all the way and sit down once without using the upper limbs. For those unable to complete the initial manoeuvre or who required assistance, the test was terminated. If successful on the initial sit to stand, participants were then asked to stand up all the way and sit down landing firmly, as fast as possible, five times without using the arms. Timing with a stopwatch was started on the command 'go' and stopped at the end of the completed fifth stand; the time taken was recorded as the participant's score.
  (1) Jones et al.
  Other Names: 5R-STS

SUMMARY:
The five-repetition sit-to-stand test has been validated and is used primarily in pulmonary medicine and cardiology, and has recently been shown to be a useful tool for the objective assessment of functional impairment in patients with degenerative diseases of the lumbar spine.

The goal of this study is to assess the possibility of supervised and unsupervised at-home-assessment. Validation of at-home-assessment would allow the 5R-STS to be easily used as a follow-up tool in clinical trials, for example.

DETAILED DESCRIPTION:
Patients will perform three 5R-STS measurements:

1. During outpatient clinics, time measured by the physician
2. At home, time measured by partner/family
3. At home, and assessed by producing a video recording of the 5R-STS performance that is subsequently sent and analyzed (time measured digitally)

ELIGIBILITY:
Inclusion Criteria:

* Degenerative diseases of the lumbar spine (Herniated disc, lumbar stenosis, spondylolisthesis, degenerative disc disease)
* Symptoms of lower back pain, neurogenic claudication, or radiculopathy

Exclusion Criteria:

* Hip or Knee prosthetics
* Walking aides

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic degenerative diseases of the lumbar spine that come in for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
5R-STS | 0 months
  Objective functional test measuring the amount of functional impairment.

SECONDARY OUTCOMES:
EQ-5D-3L | 0 months
  Validated questionnaire measuring quality of life
Oswestry Disability Index | 0 months
  Validated questionnaire measuring functional disability
VAS leg pain severity | 0 months
  Validated questionnaire measuring pain
VAS back pain severity | 0 months
  Validated questionnaire measuring pain
Roland Morris Disability Questionnaire | 0 months
  Validated questionnaire measuring functional disability

CONTACTS AND LOCATIONS:
Overall Officials: Victor E. Staartjes, MSIII, Principal Investigator — Department of Neurosurgery, Bergman Clinics, Naarden, The Netherlands
Locations (1):
- Bergman Clinics, Naarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones SE, Kon SS, Canavan JL, Patel MS, Clark AL, Nolan CM, Polkey MI, Man WD. The five-repetition sit-to-stand test as a functional outcome measure in COPD. Thorax. 2013 Nov;68(11):1015-20. doi: 10.1136/thoraxjnl-2013-203576. Epub 2013 Jun 19. PMID 23783372
- [Derived] Klukowska AM, Staartjes VE, Vandertop WP, Schroder ML. Predictors of five-repetition sit-to-stand test performance in patients with lumbar degenerative disease. Acta Neurochir (Wien). 2023 Jan;165(1):107-115. doi: 10.1007/s00701-022-05441-1. Epub 2022 Dec 7. PMID 36477416
- [Derived] Staartjes VE, Klukowska AM, Schroder ML. Association of maximum back and leg pain severity with objective functional impairment as assessed by five-repetition sit-to-stand testing: analysis of two prospective studies. Neurosurg Rev. 2020 Oct;43(5):1331-1338. doi: 10.1007/s10143-019-01168-3. Epub 2019 Aug 26. PMID 31451936
- [Derived] Staartjes VE, Beusekamp F, Schroder ML. Can objective functional impairment in lumbar degenerative disease be reliably assessed at home using the five-repetition sit-to-stand test? A prospective study. Eur Spine J. 2019 Apr;28(4):665-673. doi: 10.1007/s00586-019-05897-3. Epub 2019 Jan 24. PMID 30680635